CLINICAL TRIAL: NCT02056899
Title: Effect of Maintenance Gabapentin Therapy on the Rate of Premature Birth in Women With Preterm Labor After Receiving Tocolysis.
Brief Title: Maintenance Gabapentin to Prolong Pregnancy.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Thomas Guttuso, Associate Professor of Neurology, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 423140-2
Record Dates: First submitted 2013-07-30; First posted 2014-02-06 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Preterm Labor, Premature Birth
Keywords: Preterm labor, premature birth, gabapentin
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin
  Other Names: Neurontin

SUMMARY:
This is a pilot study to evaluate the tolerability and effects of maintenance gabapentin therapy on the rate of premature birth in women who have had preterm labor.

ELIGIBILITY:
Eligibility Criteria:

1. Healthy 18-45 year old female with singleton pregnancy, 20-34 weeks gestation, without ruptured membranes.
2. Preterm labor defined as regular uterine contractions of at least 6/hour for ≥ 1 hour with ≥ 1cm of cervical dilation or ≤ 2.5cm cervical length or any documented cervical change from the initial pelvic exam.
3. Cervical dilation not more than 4cm.
4. Initiation of a tocolytic agent (e.g. magnesium sulfate, nifedipine, indomethacin) within the previous 72 hours.
5. Pregnancy not conceived through in-vitro fertilization (IVF) due to the known higher rates of congenital defects associated with this procedure.30
6. No placenta praevia or abruptio placentae or cervical cerclage.
7. No intra-uterine growth restriction or non-reassuring fetal status.
8. No known serious fetal malformations.
9. No chorioamnionitis or medical/psychiatric/substance abuse comorbidity that may complicate the pregnancy or interfere with the subject's ability to comply with study procedures in the opinion of Dr. Guttuso or the subject's obstetrician.
10. No history of suicide attempt. No suicidal thoughts over past 6 months.
11. Not currently receiving gabapentin, pregabalin, progesterone or a known teratogenic medication and no known allergy to gabapentin therapy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Rate of premature birth (before 37 weeks gestation) | At delivery

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States